CLINICAL TRIAL: NCT04074759
Title: A Phase 1a/1b Study of FPT155 in Patients With Advanced Solid Tumors
Brief Title: FPT155 in Patients With Advanced Solid Tumors
Acronym: FPT155-001
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Five Prime Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FPT155-001
Record Dates: First submitted 2019-08-13; First posted 2019-08-30 (Actual); Results first posted 2025-01-23 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2024-02

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: Two arm trial with multiple cohorts
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FPT155 monotherapy (Experimental): The study consists of dose escalation and cohort expansions
  Interventions: Biological: FPT155
- FPT155 in combination with pembrolizumab (Experimental): The study consists of dose escalation and cohort expansions
  Interventions: Biological: FPT155; Biological: pembrolizumab

INTERVENTIONS:
Biological: FPT155 — A soluble CD80 fusion protein
Biological: pembrolizumab — An anti-PD1 antibody
  Arms: FPT155 in combination with pembrolizumab

SUMMARY:
This study is a Phase 1 open-label, first-in-human, multicenter study to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics, and activity of FPT155 as monotherapy in patients with advanced solid tumors.

DETAILED DESCRIPTION:
This Phase 1 study is comprised of dose escalation and cohort expansions for FPT155 monotherapy and for FPT155 in combination with pembrolizumab. Monotherapy dose escalation is designed with initial accelerated titration followed by a standard 3+3 dose escalation; combination dose escalation uses a standard 3+3 design. Patients will remain on study treatment until progression of disease, unacceptable toxicity, or other specified reason for discontinuation.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed solid tumors (except primary central nervous system tumors). For patients enrolled for treatment with FPT155+pembrolizumab: histologically confirmed non-small cell lung cancer not eligible for curative therapy.
* Disease that is unresectable, locally advanced, or metastatic and has progressed following all standard treatments or is not appropriate for standard treatments
* All patients must have at least one measurable lesion at baseline according to RECIST v1.1
* Availability of archival tumor tissue and consent to provide archival tumor for retrospective biomarker analysis, or consent to undergo a fresh tumor biopsy during screening
* For patients participating in cohort expansions: consent to undergo a mandatory fresh tumor biopsy during screening and on treatment
* ECOG performance status of 0 or 1
* Prior radiotherapy must be completed at least 2 weeks before first dose of study treatment administration. No radiopharmaceuticals (eg, strontium, samarium) within 8 weeks before first dose of study treatment administration.
* Prior surgery that requires general anesthesia must be completed at least 14 days before first dose of study treatment
* Adequate bone marrow, liver and kidney function

Exclusion Criteria:

* Uncontrolled or significant cardiac disease
* Any uncontrolled medical condition or psychiatric disorder including infection, autoimmune disease, bleeding disorder or symptomatic involvement of the central nervous system
* Treatment with any anti-cancer therapy or participation in another investigational drug or biologics trial within 28 days or ≤ 5 half-lives (whichever is shorter)
* Patients who discontinue prior immune-modulating therapies (including regimens containing an immune agonist or a PD-L1/PD-1 antagonist) due to toxicity or have received treatment within 5 half lives or 90 days
* Pregnancy or breastfeeding
* For patients participating in cohort expansion: Prior treatment with a CTLA-4 antagonist, including ipilimumab and tremelimumab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-10-18 (Actual); Primary Completion 2021-08-10 (Actual); Study Completion 2021-08-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (12):
- Australia (7):
  - Chris O'Brien Lifehouse, Camperdown, New South Wales
  - St Vincent's Hospital Sydney, Darlinghurst, New South Wales
  - Scientia Clinical Research, Randwick, New South Wales
  - ICON, Auchenflower, Queensland
  - Olivia Newton-John Cancer Center, Heidelberg, Victoria
  - Cabrini Hospital, Malvern, Victoria
  - Linear Clinical Research, Nedlands, Western Australia
- South Korea (5):
  - National Cancer Center, Goyang-si, Gyeonggi-do
  - St Vincent Hospital of the Catholic University of Korea, Suwon, Gyeonggi-do
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Samsung Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with advanced solid tumours were recruited across 15 centers in Australia and South Korea from October 2018 to August 2021.
Pre-assignment Details: Participants received escalating doses of FTP155 until the recommended dose (RD) was established in Phase 1a monotherapy. Phase 1b monotherapy involved dividing participants into 4 tumor-specific cohorts, treated at the RD. In Phase 1a combination therapy, participants with non-small cell lung cancer were split into 3 cohorts and given FTP155 below the RD with Pembrolizumab. Both Phase 1b monotherapy and Phase 1a combination were initiated but not completed due to the study's closure.
Groups:
- Phase 1a Monotherapy: FPT155 Dose A: Participants with advanced solid tumours received FPT155 intravenously (IV) once every 3 weeks (Q3W) in escalating doses (A-L) until the recommended dose (RD) was identified.
- Phase 1a Monotherapy: FPT155 Dose B; Phase 1a Monotherapy: FPT155 Dose C; Phase 1a Monotherapy: FPT155 Dose D; Phase 1a Monotherapy: FPT155 Dose E; Phase 1a Monotherapy: FPT155 Dose F; Phase 1a Monotherapy: FPT155 Dose G; Phase 1a Monotherapy: FPT155 Dose H; Phase 1a Monotherapy: FPT155 Dose I; Phase 1a Monotherapy: FPT155 Dose J; Phase 1a Monotherapy: FPT155 Dose K; Phase 1a Monotherapy: FPT155 Dose L: Participants with advanced solid tumours received FPT155 IV once Q3W in escalating doses (A-L) until the RD was identified.
- Phase 1b Monotherapy: 1bM1 FPT155 Dose K: Participants with advanced renal cell carcinoma were treated with FPT155 IV Q3W at the RD identified in Phase 1a monotherapy (Dose K).
- Phase 1b Monotherapy: 1bM2 FPT155 Dose K: Participants with advanced melanoma were treated with FPT155 IV Q3W at the RD identified in Phase 1a monotherapy (Dose K).
- Phase 1b Monotherapy: 1bM3 FPT155 Dose K: Participants with previously treated unresectable or metastatic non-small cell lung cancer and an absence of suitable standard treatment options were treated with FPT155 IV Q3W at the RD identified in Phase 1a monotherapy (Dose K).
- Phase 1b Monotherapy: 1bM4 FPT155 Dose K: Participants with previously treated solid tumors with a response to prior PD-1 or PDL-1 directed treatment as defined by an objective response (partial or complete response) as determined by the Investigator per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1,or a minimum of 3 months on prior PD-1 or PDL-1 directed therapy were treated with FPT155 at the RD identified in Phase 1a monotherapy (Dose K).
- Phase 1a Combination: FPT155 (Dose H) + Pembrolizumab 200 mg: Participants with non-small cell lung cancer were treated with FTB155 Dose H administered IV Q3W in combination with 200 mg Pembrolizumab.
- Phase 1a Combination: FPT155 (Dose I) + Pembrolizumab 200 mg: Participants with non-small cell lung cancer were treated with FTB155 Dose I administered IV Q3W in combination with 200 mg Pembrolizumab.
- Phase 1a Combination: FPT155 (Dose J) + Pembrolizumab 200 mg: Participants with non-small cell lung cancer were treated with FTB155 Dose J administered IV Q3W in combination with 200 mg Pembrolizumab.
Period: Overall Study
Arm/Group | Phase 1a Monotherapy: FPT155 Dose A | Phase 1a Monotherapy: FPT155 Dose B | Phase 1a Monotherapy: FPT155 Dose C | Phase 1a Monotherapy: FPT155 Dose D | Phase 1a Monotherapy: FPT155 Dose E | Phase 1a Monotherapy: FPT155 Dose F | Phase 1a Monotherapy: FPT155 Dose G | Phase 1a Monotherapy: FPT155 Dose H | Phase 1a Monotherapy: FPT155 Dose I | Phase 1a Monotherapy: FPT155 Dose J | Phase 1a Monotherapy: FPT155 Dose K | Phase 1a Monotherapy: FPT155 Dose L | Phase 1b Monotherapy: 1bM1 FPT155 Dose K | Phase 1b Monotherapy: 1bM2 FPT155 Dose K | Phase 1b Monotherapy: 1bM3 FPT155 Dose K | Phase 1b Monotherapy: 1bM4 FPT155 Dose K | Phase 1a Combination: FPT155 (Dose H) + Pembrolizumab 200 mg | Phase 1a Combination: FPT155 (Dose I) + Pembrolizumab 200 mg | Phase 1a Combination: FPT155 (Dose J) + Pembrolizumab 200 mg
Started | 1 | 1 | 2 | 1 | 4 | 3 | 3 | 3 | 7 | 10 | 20 | 6 | 1 | 5 | 3 | 1 | 3 | 3 | 3
Received at Least 1 Dose of FPT155 | 1 | 1 | 2 | 1 | 4 | 3 | 3 | 3 | 7 | 10 | 20 | 6 | 1 | 5 | 3 | 1 | 3 | 3 | 3
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 1 | 1 | 2 | 1 | 4 | 3 | 3 | 3 | 5 | 8 | 20 | 5 | 1 | 5 | 3 | 1 | 3 | 3 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 1 | 2 | 9 | 2 | 1 | 3 | 2 | 0 | 0 | 3 | 1
Not completed — Death | 1 | 0 | 1 | 1 | 2 | 0 | 1 | 0 | 3 | 2 | 4 | 1 | 0 | 2 | 1 | 0 | 1 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Not completed — Other | 0 | 1 | 1 | 0 | 2 | 1 | 2 | 1 | 1 | 4 | 4 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Missing end of study status | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population: All participants who received any portion of a least one dose of FPT155.
Groups:
- Phase 1b Monotherapy: 1bM4 FPT155 Dose K: Participants with previously treated solid tumors with a response to prior PD-1 or PDL-1 directed treatment as defined by an objective response (partial or complete response) as determined by the Investigator per RECIST v1.1,or a minimum of 3 months on prior PD-1 or PDL-1 directed therapy were treated with FPT155 at the RD identified in Phase 1a monotherapy (Dose K).
- Total: Total of all reporting groups
Arm/Group | Phase 1a Monotherapy: FPT155 Dose A | Phase 1a Monotherapy: FPT155 Dose B | Phase 1a Monotherapy: FPT155 Dose C | Phase 1a Monotherapy: FPT155 Dose D | Phase 1a Monotherapy: FPT155 Dose E | Phase 1a Monotherapy: FPT155 Dose F | Phase 1a Monotherapy: FPT155 Dose G | Phase 1a Monotherapy: FPT155 Dose H | Phase 1a Monotherapy: FPT155 Dose I | Phase 1a Monotherapy: FPT155 Dose J | Phase 1a Monotherapy: FPT155 Dose K | Phase 1a Monotherapy: FPT155 Dose L | Phase 1b Monotherapy: 1bM1 FPT155 Dose K | Phase 1b Monotherapy: 1bM2 FPT155 Dose K | Phase 1b Monotherapy: 1bM3 FPT155 Dose K | Phase 1b Monotherapy: 1bM4 FPT155 Dose K | Phase 1a Combination: FPT155 (Dose H) + Pembrolizumab 200 mg | Phase 1a Combination: FPT155 (Dose I) + Pembrolizumab 200 mg | Phase 1a Combination: FPT155 (Dose J) + Pembrolizumab 200 mg | Total
Number analyzed (Participants) | 1 | 1 | 2 | 1 | 4 | 3 | 3 | 3 | 7 | 10 | 20 | 6 | 1 | 5 | 3 | 1 | 3 | 3 | 3 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 53 (NA) — Value not estimable as only 1 participant was in the arm. | 61 (NA) — Value not estimable as only 1 participant was in the arm. | 65.5 (10.61) | 42 (NA) — Value not estimable as only 1 participant was in the arm. | 63.5 (12.61) | 64.3 (5.13) | 69 (4.58) | 53 (7.81) | 57.3 (16.55) | 58.6 (7.75) | 60.3 (12.17) | 59.3 (14.22) | 64 (NA) — Value not estimable as only 1 participant was in the arm. | 53.4 (10.33) | 64.7 (3.06) | 71 (NA) — Value not estimable as only 1 participant was in the arm. | 65.3 (3.06) | 61.0 (15.13) | 68.7 (2.52) | 60.4 (10.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 2 | 1 | 1 | 2 | 1 | 1 | 3 | 5 | 5 | 5 | 1 | 5 | 2 | 0 | 2 | 0 | 1 | 38
  Male | 0 | 1 | 0 | 0 | 3 | 1 | 2 | 2 | 4 | 5 | 15 | 1 | 0 | 0 | 1 | 1 | 1 | 3 | 2 | 42
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 4 | 12 | 1 | 1 | 5 | 3 | 0 | 0 | 3 | 1 | 33
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 1 | 1 | 2 | 1 | 4 | 3 | 3 | 2 | 3 | 5 | 7 | 5 | 0 | 0 | 0 | 1 | 3 | 0 | 2 | 43
  Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Missing | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 1 | 1 | 2 | 1 | 4 | 3 | 3 | 3 | 6 | 9 | 18 | 6 | 1 | 5 | 3 | 1 | 3 | 3 | 3 | 76
  Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
  Unknown | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced Treatment-emergent Adverse Events (TEAEs)
Description: TEAE was defined as an adverse event (AE) that was not present prior to the start date of study drug or was worsened during treatment and 100 days after last dose of treatment. An AE that was present at treatment initiation but resolved and then reappeared and the event severity increase while the participant was on treatment is also a TEAE. A severe AE (SAE) is defined as any untoward medical occurrence that at any dose: Is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, and is a congenital anomaly/birth defect. AEs were graded 1 (mild)-5 (fatal AE) according to the National Cancer Institute Common Toxicity Criteria for Adverse Events (NCI-CTCAE) Version 4.03.
Time Frame: Median (min, max) duration of FPT155 exposure was 6.57 [3.0, 49.6] weeks for the Phase 1a Monotherapy part of the study, 8.29 [3.0, 27.1] weeks for the Phase 1b Monotherapy, and 14.71 [3.0, 25.1] weeks for the Phase 1a Combination
Population: Safety population: All participants who received any portion of a least one dose of FPT155.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1a Monotherapy: FPT155 Dose A | Phase 1a Monotherapy: FPT155 Dose B | Phase 1a Monotherapy: FPT155 Dose C | Phase 1a Monotherapy: FPT155 Dose D | Phase 1a Monotherapy: FPT155 Dose E | Phase 1a Monotherapy: FPT155 Dose F | Phase 1a Monotherapy: FPT155 Dose G | Phase 1a Monotherapy: FPT155 Dose H | Phase 1a Monotherapy: FPT155 Dose I | Phase 1a Monotherapy: FPT155 Dose J | Phase 1a Monotherapy: FPT155 Dose K | Phase 1a Monotherapy: FPT155 Dose L | Phase 1b Monotherapy: 1bM1 FPT155 Dose K | Phase 1b Monotherapy: 1bM2 FPT155 Dose K | Phase 1b Monotherapy: 1bM3 FPT155 Dose K | Phase 1b Monotherapy: 1bM4 FPT155 Dose K | Phase 1a Combination: FPT155 (Dose H) + Pembrolizumab 200 mg | Phase 1a Combination: FPT155 (Dose I) + Pembrolizumab 200 mg | Phase 1a Combination: FPT155 (Dose J) + Pembrolizumab 200 mg
Number analyzed (Participants) | 1 | 1 | 2 | 1 | 4 | 3 | 3 | 3 | 7 | 10 | 20 | 6 | 1 | 5 | 3 | 1 | 3 | 3 | 3
Participants
  All TEAEs | 1 | 1 | 2 | 1 | 3 | 2 | 3 | 3 | 6 | 10 | 20 | 6 | 1 | 5 | 3 | 1 | 3 | 3 | 2
  TEAEs Grade 3 or Higher | 1 | 0 | 1 | 0 | 1 | 1 | 3 | 1 | 1 | 2 | 11 | 2 | 1 | 4 | 2 | 0 | 2 | 3 | 1
  TEAEs Related to FPT155 | 0 | 0 | 1 | 1 | 1 | 0 | 2 | 2 | 4 | 6 | 11 | 6 | 1 | 4 | 3 | 1 | 1 | 2 | 2
  All SAEs | 1 | 0 | 1 | 0 | 1 | 1 | 3 | 0 | 2 | 3 | 10 | 2 | 1 | 0 | 2 | 0 | 2 | 3 | 2
  SAEs Related to FPT155 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 0 | 0 | 2 | 0 | 0 | 0 | 2
  TEAEs Leading to Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Phase 1a Monotherapy: Number of Participants Who Experienced Dose Limiting Toxicities (DLTs)
Description: DLTs ware defined as any of the events that occurred during the first 28 days of treatment and were assessed by the Clinical Research Coordinator (CRC) as related to FPT155.
Time Frame: Cycle 1 (one cycle = 21 days) Day 1 post-dose, up to approximately 21 days
Population: DLT-evaluable population: All participants enrolled into Phase 1a dose escalation portion of the study who received at least 1 dose of all assigned study drug(s) and remain on study for the 21-day DLT evaluation period, or who experienced a DLT before clearing the 21-day DLT evaluation interval. Study used a 3 + 3 design in the Phase 1a Monotherapy cohorts, from cohort "Phase 1a Monotherapy: FPT155 Dose E".
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1a Monotherapy: FPT155 Dose A | Phase 1a Monotherapy: FPT155 Dose B | Phase 1a Monotherapy: FPT155 Dose C | Phase 1a Monotherapy: FPT155 Dose D | Phase 1a Monotherapy: FPT155 Dose E | Phase 1a Monotherapy: FPT155 Dose F | Phase 1a Monotherapy: FPT155 Dose G | Phase 1a Monotherapy: FPT155 Dose H | Phase 1a Monotherapy: FPT155 Dose I | Phase 1a Monotherapy: FPT155 Dose J | Phase 1a Monotherapy: FPT155 Dose K | Phase 1a Monotherapy: FPT155 Dose L
Number analyzed (Participants) | 1 | 1 | 2 | 1 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 6
Participants
  All DLTs | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Cytokine release syndrome | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Infusion related reaction | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

3. Primary Outcome: Phase 1b Monotherapy: Number of Participants Who Had FPT155 Treatment Discontinued Due to AEs
Description: Represents the number of participants who had discontinuation of FPT155 dosing due to AEs.
Time Frame: Median (min, max) duration of FPT155 exposure was 8.29 [3.0, 27.1] weeks.
Population: Safety population: All participants who received any portion of a least one dose of FPT155.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b Monotherapy: 1bM1 FPT155 Dose K | Phase 1b Monotherapy: 1bM2 FPT155 Dose K | Phase 1b Monotherapy: 1bM3 FPT155 Dose K | Phase 1b Monotherapy: 1bM4 FPT155 Dose K
Number analyzed (Participants) | 1 | 5 | 3 | 1
Participants | 0 | 0 | 2 | 0

4. Primary Outcome: Phase 1b Monotherapy: Number of Participants Who Had FPT155 Treatment Modified Due to AEs
Description: Represents the number of participants who had a modification in the dosing schedules of FPT155 due to AEs.
Time Frame: Median (min, max) duration of FPT155 exposure was 8.29 [3.0, 27.1] weeks.
Population: Safety population: All participants who received any portion of a least one dose of FPT155.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b Monotherapy: 1bM1 FPT155 Dose K | Phase 1b Monotherapy: 1bM2 FPT155 Dose K | Phase 1b Monotherapy: 1bM3 FPT155 Dose K | Phase 1b Monotherapy: 1bM4 FPT155 Dose K
Number analyzed (Participants) | 1 | 5 | 3 | 1
Participants | 0 | 1 | 0 | 0

5. Primary Outcome: Phase 1b Monotherapy: Number of Participants Who Had FPT155 Treatment Interrupted Due to AEs
Description: Represents the number of participants who had an interruption in the dosing schedules of FPT155 due to AEs.
Time Frame: Median (min, max) duration of FPT155 exposure was 8.29 [3.0, 27.1] weeks.
Population: Safety population: All participants who received any portion of a least one dose of FPT155.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b Monotherapy: 1bM1 FPT155 Dose K | Phase 1b Monotherapy: 1bM2 FPT155 Dose K | Phase 1b Monotherapy: 1bM3 FPT155 Dose K | Phase 1b Monotherapy: 1bM4 FPT155 Dose K
Number analyzed (Participants) | 1 | 5 | 3 | 1
Participants | 0 | 1 | 0 | 0

6. Primary Outcome: Phase 1a Combination: Number of Participants Who Experienced DLTs
Description: DLTs ware defined as any of the events that occur during the first 28 days of treatment and are assessed by the CRC as related to FPT155.
Time Frame: Cycle 1 (one cycle = 21 days) Day 1 post-dose, up to approximately 21 days
Population: DLT-evaluable population: All participants enrolled into Phase 1a dose escalation portion of the study who received at least 1 dose of all assigned study drug(s) and remain on study for the 21-day DLT evaluation period, or who experienced a DLT before clearing the 21-day DLT evaluation interval.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1a Combination: FPT155 (Dose H) + Pembrolizumab 200 mg | Phase 1a Combination: FPT155 (Dose I) + Pembrolizumab 200 mg | Phase 1a Combination: FPT155 (Dose J) + Pembrolizumab 200 mg
Number analyzed (Participants) | 3 | 3 | 3
Participants
  All DLTs | 0 | 0 | 1
  Cytokine release syndrome | 0 | 0 | 1
  Aspartate aminotransferase increased | 0 | 0 | 1

7. Secondary Outcome: Phase 1a Monotherapy: Area Under Serum Concentration-time Profile From Time 0 to Time Tau (The Dosing Interval) (AUC0-tau) of FPT155
Time Frame: Cycle 1 (21-day cycles) Day 1 pre-dose, Day 1 (15min, 1h, 2h, 6h post-dose), Day 2, Day 4, Day 8, Day 15
Population: PK-Evaluable Population: All participants who received at least one dose of study drug, and had sufficient PK sample for the calculation of at least one PK parameter on at least one Study Day, and had evaluable data.
Measure: Mean (Standard Deviation); unit: day*ug/mL
Groups:
- Phase 1a Monotherapy: FPT155 Dose A; Phase 1a Monotherapy: FPT155 Dose B; Phase 1a Monotherapy: FPT155 Dose C; Phase 1a Monotherapy: FPT155 Dose D; Phase 1a Monotherapy: FPT155 Dose E; Phase 1a Monotherapy: FPT155 Dose F; Phase 1a Monotherapy: FPT155 Dose G; Phase 1a Monotherapy: FPT155 Dose H; Phase 1a Monotherapy: FPT155 Dose I; Phase 1a Monotherapy: FPT155 Dose J; Phase 1a Monotherapy: FPT155 Dose K; Phase 1a Monotherapy: FPT155 Dose L: Participants with advanced solid tumours received FPT155 IV once Q3W in escalating doses (A-L) until the RD was identified.
Arm/Group | Phase 1a Monotherapy: FPT155 Dose A | Phase 1a Monotherapy: FPT155 Dose B | Phase 1a Monotherapy: FPT155 Dose C | Phase 1a Monotherapy: FPT155 Dose D | Phase 1a Monotherapy: FPT155 Dose E | Phase 1a Monotherapy: FPT155 Dose F | Phase 1a Monotherapy: FPT155 Dose G | Phase 1a Monotherapy: FPT155 Dose H | Phase 1a Monotherapy: FPT155 Dose I | Phase 1a Monotherapy: FPT155 Dose J | Phase 1a Monotherapy: FPT155 Dose K | Phase 1a Monotherapy: FPT155 Dose L
Number analyzed (Participants) | 1 | 1 | 2 | 1 | 4 | 3 | 3 | 3 | 7 | 10 | 16 | 2
day*ug/mL | 0.0327 (NA) — Value not estimable as only 1 participant was in the arm. | 0.1586 (NA) — Value not estimable as only 1 participant was in the arm. | 1.1365 (0.36220) | 2.4057 (NA) — Value not estimable as only 1 participant was in the arm. | 7.6030 (1.70572) | 20.9191 (2.58340) | 38.4803 (5.39054) | 73.3365 (20.47867) | 165.9985 (38.97415) | 318.4115 (55.46423) | 680.4735 (186.74665) | 578.2617 (411.33336)

8. Secondary Outcome: Phase 1a Monotherapy: Maximum Observed Serum Concentration (Cmax) of FPT155
Time Frame: Cycle 1 (21-day cycles) Day 1 pre-dose, Day 1 (15min, 1h, 2h, 6h post-dose), Day 2, Day 4, Day 8, Day 15
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Phase 1a Monotherapy: FPT155 Dose A | Phase 1a Monotherapy: FPT155 Dose B | Phase 1a Monotherapy: FPT155 Dose C | Phase 1a Monotherapy: FPT155 Dose D | Phase 1a Monotherapy: FPT155 Dose E | Phase 1a Monotherapy: FPT155 Dose F | Phase 1a Monotherapy: FPT155 Dose G | Phase 1a Monotherapy: FPT155 Dose H | Phase 1a Monotherapy: FPT155 Dose I | Phase 1a Monotherapy: FPT155 Dose J | Phase 1a Monotherapy: FPT155 Dose K | Phase 1a Monotherapy: FPT155 Dose L
Number analyzed (Participants) | 1 | 1 | 2 | 1 | 4 | 3 | 3 | 3 | 7 | 10 | 17 | 2
ug/mL | 0.0152 (NA) — Value not estimable as only 1 participant was in the arm. | 0.0398 (NA) — Value not estimable as only 1 participant was in the arm. | 0.3185 (0.19304) | 0.4440 (NA) — Value not estimable as only 1 participant was in the arm. | 1.7033 (0.37909) | 4.1403 (1.00748) | 8.2337 (0.99910) | 15.0070 (1.67983) | 42.4436 (14.15113) | 74.4304 (12.04634) | 154.4599 (36.68364) | 236.0270 (91.32991)

9. Secondary Outcome: Phase 1a Monotherapy: Trough Observed Serum Concentration at the End of Each Dose Interval (Ctrough) of FPT155
Time Frame: Cycle 1 (21-day cycles) Day 1 pre-dose, Day 1 (15min, 1h, 2h, 6h post-dose), Day 2, Day 4, Day 8, Day 15
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Phase 1a Monotherapy: FPT155 Dose A | Phase 1a Monotherapy: FPT155 Dose B | Phase 1a Monotherapy: FPT155 Dose C | Phase 1a Monotherapy: FPT155 Dose D | Phase 1a Monotherapy: FPT155 Dose E | Phase 1a Monotherapy: FPT155 Dose F | Phase 1a Monotherapy: FPT155 Dose G | Phase 1a Monotherapy: FPT155 Dose H | Phase 1a Monotherapy: FPT155 Dose I | Phase 1a Monotherapy: FPT155 Dose J | Phase 1a Monotherapy: FPT155 Dose K | Phase 1a Monotherapy: FPT155 Dose L
Number analyzed (Participants) | 0 | 0 | 1 | 1 | 4 | 3 | 3 | 3 | 7 | 9 | 12 | 1
ug/mL |  |  | 0.0097 (NA) — Value not estimable as only 1 participant was in the arm. | 0.0211 (NA) — Value not estimable as only 1 participant was in the arm. | 0.0670 (0.03697) | 0.2827 (0.02203) | 0.2793 (0.02875) | 0.9813 (0.72419) | 1.8921 (0.97118) | 3.0308 (0.97789) | 8.1734 (3.79640) | 8.0930 (NA) — Value not estimable as only 1 participant was in the arm.

10. Secondary Outcome: Phase 1a Monotherapy: Clearance (CL) of FPT155
Time Frame: Cycle 1 (21-day cycles) Day 1 pre-dose, Day 1 (15min, 1h, 2h, 6h post-dose), Day 2, Day 4, Day 8, Day 15
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mL/day
Arm/Group | Phase 1a Monotherapy: FPT155 Dose A | Phase 1a Monotherapy: FPT155 Dose B | Phase 1a Monotherapy: FPT155 Dose C | Phase 1a Monotherapy: FPT155 Dose D | Phase 1a Monotherapy: FPT155 Dose E | Phase 1a Monotherapy: FPT155 Dose F | Phase 1a Monotherapy: FPT155 Dose G | Phase 1a Monotherapy: FPT155 Dose H | Phase 1a Monotherapy: FPT155 Dose I | Phase 1a Monotherapy: FPT155 Dose J | Phase 1a Monotherapy: FPT155 Dose K | Phase 1a Monotherapy: FPT155 Dose L
Number analyzed (Participants) | 0 | 0 | 1 | 1 | 4 | 3 | 3 | 3 | 7 | 10 | 13 | 1
mL/day |  |  | 723.1295 (NA) — Value not estimable as only 1 participant was in the arm. | 816.5143 (NA) — Value not estimable as only 1 participant was in the arm. | 872.7624 (177.16607) | 885.2506 (121.93486) | 1023.0799 (117.05581) | 921.2589 (387.65387) | 803.7378 (247.88188) | 838.7004 (152.86047) | 822.2251 (308.79493) | 893.7646 (NA) — Value not estimable as only 1 participant was in the arm.

11. Secondary Outcome: Phase 1a Monotherapy: Terminal Half-life (t1/2) of FPT155
Time Frame: Cycle 1 (21-day cycles) Day 1 pre-dose, Day 1 (15min, 1h, 2h, 6h post-dose), Day 2, Day 4, Day 8, Day 15
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Phase 1a Monotherapy: FPT155 Dose A | Phase 1a Monotherapy: FPT155 Dose B | Phase 1a Monotherapy: FPT155 Dose C | Phase 1a Monotherapy: FPT155 Dose D | Phase 1a Monotherapy: FPT155 Dose E | Phase 1a Monotherapy: FPT155 Dose F | Phase 1a Monotherapy: FPT155 Dose G | Phase 1a Monotherapy: FPT155 Dose H | Phase 1a Monotherapy: FPT155 Dose I | Phase 1a Monotherapy: FPT155 Dose J | Phase 1a Monotherapy: FPT155 Dose K | Phase 1a Monotherapy: FPT155 Dose L
Number analyzed (Participants) | 0 | 0 | 1 | 1 | 4 | 3 | 3 | 3 | 7 | 10 | 13 | 1
hours |  |  | 6.2328 (NA) — Value not estimable as only 1 participant was in the arm. | 5.5142 (NA) — Value not estimable as only 1 participant was in the arm. | 6.2067 (0.61062) | 7.5696 (0.69887) | 5.3969 (0.40483) | 6.7752 (2.32987) | 6.9751 (1.62270) | 5.8128 (0.80921) | 5.9846 (1.27669) | 5.3674 (NA) — Value not estimable as only 1 participant was in the arm.

12. Secondary Outcome: Phase 1a Monotherapy: Volume of Distribution at Steady State (Vss) of FPT155
Time Frame: Cycle 1 (21-day cycles) Day 1 pre-dose, Day 1 (15min, 1h, 2h, 6h post-dose), Day 2, Day 4, Day 8, Day 15
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Phase 1a Monotherapy: FPT155 Dose A | Phase 1a Monotherapy: FPT155 Dose B | Phase 1a Monotherapy: FPT155 Dose C | Phase 1a Monotherapy: FPT155 Dose D | Phase 1a Monotherapy: FPT155 Dose E | Phase 1a Monotherapy: FPT155 Dose F | Phase 1a Monotherapy: FPT155 Dose G | Phase 1a Monotherapy: FPT155 Dose H | Phase 1a Monotherapy: FPT155 Dose I | Phase 1a Monotherapy: FPT155 Dose J | Phase 1a Monotherapy: FPT155 Dose K | Phase 1a Monotherapy: FPT155 Dose L
Number analyzed (Participants) | 0 | 0 | 1 | 1 | 4 | 3 | 3 | 3 | 7 | 10 | 13 | 1
mL |  |  | 5589.3077 (NA) — Value not estimable as only 1 participant was in the arm. | 5945.0963 (NA) — Value not estimable as only 1 participant was in the arm. | 6390.4335 (974.58304) | 8258.2000 (1221.67174) | 7073.7877 (1555.88613) | 6994.1331 (672.03487) | 6413.4280 (1007.47809) | 5958.4609 (1409.10784) | 5945.5205 (1442.85088) | 6032.9646 (NA) — Value not estimable as only 1 participant was in the arm.

13. Secondary Outcome: Phase 1a Monotherapy: Number of Participants With Treatment-emergent Anti-FPT155 Antibody Response
Description: Data presented below includes participants with at least 1 anti-drug antibodies-positive sample relative to baseline after initiation of the treatment.
Time Frame: Cycle 1 (21-day cycles) Day 1
Population: Safety population: All participants who received any portion of a least one dose of FPT155.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1a Monotherapy: FPT155 Dose A | Phase 1a Monotherapy: FPT155 Dose B | Phase 1a Monotherapy: FPT155 Dose C | Phase 1a Monotherapy: FPT155 Dose D | Phase 1a Monotherapy: FPT155 Dose E | Phase 1a Monotherapy: FPT155 Dose F | Phase 1a Monotherapy: FPT155 Dose G | Phase 1a Monotherapy: FPT155 Dose H | Phase 1a Monotherapy: FPT155 Dose I | Phase 1a Monotherapy: FPT155 Dose J | Phase 1a Monotherapy: FPT155 Dose K | Phase 1a Monotherapy: FPT155 Dose L
Number analyzed (Participants) | 1 | 1 | 2 | 1 | 4 | 3 | 3 | 3 | 7 | 10 | 20 | 6
Participants
  Anti-FPT155 Positive | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 3 | 1 | 3 | 0
  Anti-FPT155 Negative | 1 | 1 | 2 | 1 | 3 | 1 | 3 | 2 | 4 | 8 | 9 | 0
  Not Evaluable | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 8 | 6

14. Secondary Outcome: Phase 1b Monotherapy: Objective Response Rate (ORR) Per RECIST v1.1
Description: ORR was defined as the total number of participants with confirmed responses of either complete response (CR) (CR: The disappearance of all target lesions, any pathological lymph nodes [whether target or non-target] must have a reduction in short axis to <10 mm) or partial response (PR) (PR: At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters), as determined by the investigator per RECIST v1.1.
Time Frame: Up to approximately 30 months
Population: Efficacy Population: All participants who received any portion of at least one dose of FPT155.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b Monotherapy: 1bM1 FPT155 Dose K | Phase 1b Monotherapy: 1bM2 FPT155 Dose K | Phase 1b Monotherapy: 1bM3 FPT155 Dose K | Phase 1b Monotherapy: 1bM4 FPT155 Dose K
Number analyzed (Participants) | 1 | 5 | 3 | 1
Participants | 0 | 0 | 0 | 0

15. Secondary Outcome: Phase 1b Monotherapy: Duration of Response (DOR) Per RECIST v1.1
Description: DOR was defined as the time from first response (CR [The disappearance of all target lesions, any pathological lymph nodes {whether target or non-target} or PR [At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters] determined by the investigator per RECIST v1.1) that was subsequently confirmed until the onset of progressive disease (DP) (DP: At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study [this includes the baseline sum if that is the smallest on study]. In addition to the 20% relative increase, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered progression) or death from any cause, whichever occurred first.
Time Frame: Up to approximately 30 months
Population: Efficacy population inclusive of participants with CR or PR.
Arm/Group | Phase 1b Monotherapy: 1bM1 FPT155 Dose K | Phase 1b Monotherapy: 1bM2 FPT155 Dose K | Phase 1b Monotherapy: 1bM3 FPT155 Dose K | Phase 1b Monotherapy: 1bM4 FPT155 Dose K
Number analyzed (Participants) | 0 | 0 | 0 | 0

16. Secondary Outcome: Phase 1b Monotherapy: Progression-free Survival (PFS) Per RECIST v1.1
Description: PFS was defined as time from the first dose of study treatment until the first documentation by the investigator of DP (DP: At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study [this includes the baseline sum if that is the smallest on study]. In addition to the 20% relative increase, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered progression) per RECIST v1.1 or death from any cause, whichever occurred first. The median was estimated by using the Kaplan-Meier method and corresponding 2-sided 90% CI using Brookmeyer and Crowley methodology.
Time Frame: Up to approximately 30 months
Population: Efficacy Population: All participants who received any portion of at least one dose of FPT155.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Phase 1b Monotherapy: 1bM1 FPT155 Dose K | Phase 1b Monotherapy: 1bM2 FPT155 Dose K | Phase 1b Monotherapy: 1bM3 FPT155 Dose K | Phase 1b Monotherapy: 1bM4 FPT155 Dose K
Number analyzed (Participants) | 1 | 5 | 3 | 1
months | 1.31 [NA to NA] — Due to the low number of participants (1) there are too few observations (1) that impacted the estimate of the survival function to no variation, hence the 90% CIs could not be estimated. | 1.38 [0.72 to 5.42] | 4.01 [1.18 to NA] — Upper CI could not be calculated due to the low number of observations. | 1.41 [NA to NA] — Due to the low number of participants (1) there are too few observations (1) that impacted the estimate of the survival function to no variation, hence the 90% CIs could not be estimated.

17. Secondary Outcome: Phase 1b Monotherapy: Disease Control Rate (DCR) Per RECIST v1.1
Description: DCR was defined as the total number of participants with confirmed responses of either CR (CR: The disappearance of all target lesions, any pathological lymph nodes [whether target or non-target] must have a reduction in short axis to <10 mm), PR (PR: At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters), or stable disease (SD) (SD: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD. In numerical terms, it means a reduction in tumor size that is less than 30% [which is required for PR] and an increase in size that is less than 20% [which is required for PD]) as determined by the investigator per RECIST v1.1.
Time Frame: Up to approximately 30 months
Population: Efficacy Population: All participants who received any portion of at least one dose of FPT155.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b Monotherapy: 1bM1 FPT155 Dose K | Phase 1b Monotherapy: 1bM2 FPT155 Dose K | Phase 1b Monotherapy: 1bM3 FPT155 Dose K | Phase 1b Monotherapy: 1bM4 FPT155 Dose K
Number analyzed (Participants) | 1 | 5 | 3 | 1
Participants | 0 | 2 | 2 | 0

18. Secondary Outcome: Phase 1b Monotherapy: AUC0-tau of FPT155
Time Frame: Cycle 1 (21-day cycles) Day 1 pre-dose, Day 1 (15min, 1h, 2h, 6h post-dose), Day 2, Day 4, Day 8, Day 15
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: day*ug/mL
Arm/Group | Phase 1b Monotherapy: 1bM1 FPT155 Dose K | Phase 1b Monotherapy: 1bM2 FPT155 Dose K | Phase 1b Monotherapy: 1bM3 FPT155 Dose K | Phase 1b Monotherapy: 1bM4 FPT155 Dose K
Number analyzed (Participants) | 1 | 4 | 3 | 1
day*ug/mL | 785.6775 (NA) — Value not estimable as only 1 participant was in the arm. | 874.0402 (236.97475) | 827.3523 (314.06602) | 245.5924 (NA) — Value not estimable as only 1 participant was in the arm.

19. Secondary Outcome: Phase 1b Monotherapy: Cmax of FPT155
Time Frame: Cycle 1 (21-day cycles) Day 1 pre-dose, Day 1 (15min, 1h, 2h, 6h post-dose), Day 2, Day 4, Day 8, Day 15
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Phase 1b Monotherapy: 1bM1 FPT155 Dose K | Phase 1b Monotherapy: 1bM2 FPT155 Dose K | Phase 1b Monotherapy: 1bM3 FPT155 Dose K | Phase 1b Monotherapy: 1bM4 FPT155 Dose K
Number analyzed (Participants) | 1 | 4 | 3 | 1
ug/mL | 203.4790 (NA) — Value not estimable as only 1 participant was in the arm. | 180.9630 (51.85915) | 214.5727 (86.57029) | 178.5870 (NA) — Value not estimable as only 1 participant was in the arm.

20. Secondary Outcome: Phase 1b Monotherapy: Ctrough of FPT155
Time Frame: Cycle 1 (21-day cycles) Day 1 pre-dose, Day 1 (15min, 1h, 2h, 6h post-dose), Day 2, Day 4, Day 8, Day 15
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Phase 1b Monotherapy: 1bM1 FPT155 Dose K | Phase 1b Monotherapy: 1bM2 FPT155 Dose K | Phase 1b Monotherapy: 1bM3 FPT155 Dose K | Phase 1b Monotherapy: 1bM4 FPT155 Dose K
Number analyzed (Participants) | 1 | 2 | 2 | 0
ug/mL | 1.2920 (NA) — Value not estimable as only 1 participant was in the arm. | 11.6875 (0.77428) | 5.5480 (0.58266) |

21. Secondary Outcome: Phase 1b Monotherapy: CL of FPT155
Time Frame: Cycle 1 (21-day cycles) Day 1 pre-dose, Day 1 (15min, 1h, 2h, 6h post-dose), Day 2, Day 4, Day 8, Day 15
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mL/day
Arm/Group | Phase 1b Monotherapy: 1bM1 FPT155 Dose K | Phase 1b Monotherapy: 1bM2 FPT155 Dose K | Phase 1b Monotherapy: 1bM3 FPT155 Dose K | Phase 1b Monotherapy: 1bM4 FPT155 Dose K
Number analyzed (Participants) | 1 | 3 | 3 | 0
mL/day | 662.0429 (NA) — Value not estimable as only 1 participant was in the arm. | 555.8419 (119.27137) | 698.3282 (278.39932) |

22. Secondary Outcome: Phase 1b Monotherapy: t1/2 of FPT155
Time Frame: Cycle 1 (21-day cycles) Day 1 pre-dose, Day 1 (15min, 1h, 2h, 6h post-dose), Day 2, Day 4, Day 8, Day 15
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: day
Arm/Group | Phase 1b Monotherapy: 1bM1 FPT155 Dose K | Phase 1b Monotherapy: 1bM2 FPT155 Dose K | Phase 1b Monotherapy: 1bM3 FPT155 Dose K | Phase 1b Monotherapy: 1bM4 FPT155 Dose K
Number analyzed (Participants) | 1 | 3 | 3 | 0
day | 5.7318 (NA) — Value not estimable as only 1 participant was in the arm. | 6.9369 (1.38733) | 5.7844 (0.33807) |

23. Secondary Outcome: Phase 1b Monotherapy: Vss of FPT155
Time Frame: Cycle 1 (21-day cycles) Day 1 pre-dose, Day 1 (15min, 1h, 2h, 6h post-dose), Day 2, Day 4, Day 8, Day 15
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Phase 1b Monotherapy: 1bM1 FPT155 Dose K | Phase 1b Monotherapy: 1bM2 FPT155 Dose K | Phase 1b Monotherapy: 1bM3 FPT155 Dose K | Phase 1b Monotherapy: 1bM4 FPT155 Dose K
Number analyzed (Participants) | 1 | 3 | 3 | 0
mL | 3492.6594 (NA) — Value not estimable as only 1 participant was in the arm. | 5006.6203 (1687.10134) | 4934.4888 (1711.72574) |

24. Secondary Outcome: Phase 1b Monotherapy: Number of Participants With Treatment-emergent Anti-FPT155 Antibody Response
Description: as for outcome 13
Time Frame: Cycle 1 (21-day cycles) Day 1
Population: Safety population: All participants who received any portion of a least one dose of FPT155.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b Monotherapy: 1bM1 FPT155 Dose K | Phase 1b Monotherapy: 1bM2 FPT155 Dose K | Phase 1b Monotherapy: 1bM3 FPT155 Dose K | Phase 1b Monotherapy: 1bM4 FPT155 Dose K
Number analyzed (Participants) | 1 | 5 | 3 | 1
Participants
  Anti-FPT155 Positive | 0 | 0 | 0 | 0
  Anti-FPT155 Negative | 0 | 2 | 3 | 0
  Not Evaluable | 1 | 3 | 0 | 1

25. Secondary Outcome: Phase 1a Combination: ORR Per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
Description: ORR was defined as the total number of participants with confirmed responses of either CR (CR: The disappearance of all target lesions, any pathological lymph nodes [whether target or non-target] must have a reduction in short axis to <10 mm) or PR (PR: At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters), as determined by the investigator per RECIST v1.1.
Time Frame: Up to approximately 30 months
Population: Efficacy Population: All participants who received any portion of at least one dose of FPT155.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1a Combination: FPT155 (Dose H) + Pembrolizumab 200 mg | Phase 1a Combination: FPT155 (Dose I) + Pembrolizumab 200 mg | Phase 1a Combination: FPT155 (Dose J) + Pembrolizumab 200 mg
Number analyzed (Participants) | 3 | 3 | 3
Participants | 0 | 1 | 0

ADVERSE EVENTS:
Time Frame: Median (min, max) duration of FPT155 exposure was 6.57 [3.0, 49.6] weeks for the Phase 1a Monotherapy part of the study, 8.29 [3.0, 27.1] weeks for the Phase 1b Monotherapy, and 14.71 [3.0, 25.1] weeks for the Phase 1a Combination. Time frame for all-cause mortality was up to approximately 30 months.
Description: A TEAE is an AE not present before the study drug or worsened during treatment and within 100 days after the last dose. An SAE is any untoward medical occurrence that is life-threatening, requires hospitalization or prolongs it, results in persistent disability/incapacity, or is a congenital anomaly/birth defect.
Groups:
- Phase 1a Monotherapy: FPT155 Dose A: Participants with advanced solid tumours received FPT155 IV Q3W in escalating doses (A-L) until the RD was identified.
Arm/Group | Phase 1a Monotherapy: FPT155 Dose A | Phase 1a Monotherapy: FPT155 Dose B | Phase 1a Monotherapy: FPT155 Dose C | Phase 1a Monotherapy: FPT155 Dose D | Phase 1a Monotherapy: FPT155 Dose E | Phase 1a Monotherapy: FPT155 Dose F | Phase 1a Monotherapy: FPT155 Dose G | Phase 1a Monotherapy: FPT155 Dose H | Phase 1a Monotherapy: FPT155 Dose I | Phase 1a Monotherapy: FPT155 Dose J | Phase 1a Monotherapy: FPT155 Dose K | Phase 1a Monotherapy: FPT155 Dose L | Phase 1b Monotherapy: 1bM1 FPT155 Dose K | Phase 1b Monotherapy: 1bM2 FPT155 Dose K | Phase 1b Monotherapy: 1bM3 FPT155 Dose K | Phase 1b Monotherapy: 1bM4 FPT155 Dose K | Phase 1a Combination: FPT155 (Dose H) + Pembrolizumab 200 mg | Phase 1a Combination: FPT155 (Dose I) + Pembrolizumab 200 mg | Phase 1a Combination: FPT155 (Dose J) + Pembrolizumab 200 mg
All-Cause Mortality (participants affected / at risk) | 1/1 | 0/1 | 1/2 | 1/1 | 2/4 | 0/3 | 1/3 | 0/3 | 3/7 | 2/10 | 4/20 | 1/6 | 0/1 | 2/5 | 1/3 | 0/1 | 1/3 | 0/3 | 1/3
Serious Adverse Events (participants affected / at risk) | 1/1 | 0/1 | 1/2 | 0/1 | 1/4 | 1/3 | 3/3 | 0/3 | 2/7 | 3/10 | 10/20 | 2/6 | 1/1 | 0/5 | 2/3 | 0/1 | 2/3 | 3/3 | 2/3
Other Adverse Events (participants affected / at risk) | 0/1 | 1/1 | 2/2 | 1/1 | 3/4 | 2/3 | 3/3 | 3/3 | 6/7 | 10/10 | 18/20 | 5/6 | 1/1 | 5/5 | 3/3 | 1/1 | 3/3 | 3/3 | 2/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1a Monotherapy: FPT155 Dose A (N=1) | Phase 1a Monotherapy: FPT155 Dose B (N=1) | Phase 1a Monotherapy: FPT155 Dose C (N=2) | Phase 1a Monotherapy: FPT155 Dose D (N=1) | Phase 1a Monotherapy: FPT155 Dose E (N=4) | Phase 1a Monotherapy: FPT155 Dose F (N=3) | Phase 1a Monotherapy: FPT155 Dose G (N=3) | Phase 1a Monotherapy: FPT155 Dose H (N=3) | Phase 1a Monotherapy: FPT155 Dose I (N=7) | Phase 1a Monotherapy: FPT155 Dose J (N=10) | Phase 1a Monotherapy: FPT155 Dose K (N=20) | Phase 1a Monotherapy: FPT155 Dose L (N=6) | Phase 1b Monotherapy: 1bM1 FPT155 Dose K (N=1) | Phase 1b Monotherapy: 1bM2 FPT155 Dose K (N=5) | Phase 1b Monotherapy: 1bM3 FPT155 Dose K (N=3) | Phase 1b Monotherapy: 1bM4 FPT155 Dose K (N=1) | Phase 1a Combination: FPT155 (Dose H) + Pembrolizumab 200 mg (N=3) | Phase 1a Combination: FPT155 (Dose I) + Pembrolizumab 200 mg (N=3) | Phase 1a Combination: FPT155 (Dose J) + Pembrolizumab 200 mg (N=3)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Suprapubic pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Biliary obstruction (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Immune-mediated hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypophagia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Central nervous system lesion (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hemiparesis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Polyneuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Giant cell arteritis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1a Monotherapy: FPT155 Dose A (N=1) | Phase 1a Monotherapy: FPT155 Dose B (N=1) | Phase 1a Monotherapy: FPT155 Dose C (N=2) | Phase 1a Monotherapy: FPT155 Dose D (N=1) | Phase 1a Monotherapy: FPT155 Dose E (N=4) | Phase 1a Monotherapy: FPT155 Dose F (N=3) | Phase 1a Monotherapy: FPT155 Dose G (N=3) | Phase 1a Monotherapy: FPT155 Dose H (N=3) | Phase 1a Monotherapy: FPT155 Dose I (N=7) | Phase 1a Monotherapy: FPT155 Dose J (N=10) | Phase 1a Monotherapy: FPT155 Dose K (N=20) | Phase 1a Monotherapy: FPT155 Dose L (N=6) | Phase 1b Monotherapy: 1bM1 FPT155 Dose K (N=1) | Phase 1b Monotherapy: 1bM2 FPT155 Dose K (N=5) | Phase 1b Monotherapy: 1bM3 FPT155 Dose K (N=3) | Phase 1b Monotherapy: 1bM4 FPT155 Dose K (N=1) | Phase 1a Combination: FPT155 (Dose H) + Pembrolizumab 200 mg (N=3) | Phase 1a Combination: FPT155 (Dose I) + Pembrolizumab 200 mg (N=3) | Phase 1a Combination: FPT155 (Dose J) + Pembrolizumab 200 mg (N=3)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 3 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Visual acuity reduced (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 4 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 3 | 2 | 1 | 0 | 1 | 0 | 0 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 4 | 3 | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Catheter site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 2 | 1 | 1 | 2 | 3 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Feeling cold (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infusion site reaction (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Escherichia sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Otitis media acute (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Transaminases increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 3 | 3 | 0 | 0 | 1 | 0 | 0 | 2 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fluid retention (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ataxia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lumbosacral radiculopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Breast pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cold sweat (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 4 | 4 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphoedema (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Phlebitis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Venous occlusion (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-09-14): https://cdn.clinicaltrials.gov/large-docs/59/NCT04074759/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-17): https://cdn.clinicaltrials.gov/large-docs/59/NCT04074759/SAP_001.pdf